CLINICAL TRIAL: NCT04929197
Title: Evaluation of the Feasibility of Developing Personalized Breast Cancer Radiotherapy Assistive Device With Three-dimensional Printing Secondary IDs:
Brief Title: Evaluation of the Feasibility of Developing Personalized Breast Cancer Radiotherapy Assistive Device With 3D Printing
Acronym: PERSBRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N201603037
Record Dates: First submitted 2021-05-31; First posted 2021-06-18 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Breast Neoplasms; Breast Cancer; Left Sided Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Unilateral Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wear Personalized breast holder system (PERSBRA) to receiving radiotherapy (Experimental): Wear PERSBRA to the end of radiotherapy.
  Interventions: Device: PERSBRA

INTERVENTIONS:
Device: PERSBRA — After the patient is in the semi-prone position, the body shape and breast position images are obtained by the stereo scanning technology, and then using 3d printing technology to print PERSBRA.
  PERSBRA maintain a favorable new breast position in the supine position during routine radiotherapy, the cardiopulmonary dose during radiotherapy can be reduced by wearing PERSBRA.

SUMMARY:
Breast cancer is the most common malignancy among women worldwide. For early stage breast cancer, adjuvant radiotherapy is essential to minimize loco-regional disease recurrence. However, significant portions of the heart and the lungs are exposed to low dose radiation during radiotherapy, which result in stochastic side effects among breast cancer survivors. Inspired by 3D printing technology, we approached this issue with an in-house made PERSonalized BReAst holder system (PERSBRA). PERSBRA is composed of a 3D-printed plastic holder covering the whole breast and an air-filled interface. Its main function is to reproducibly adjust the breast position to decrease heart and lung radiation exposure in tangential fields. Here we propose to measure the performance of PERSBR in terms of radiation dosimetry in 50 patients receiving scheduled whole breast irradiation. For customized PERSBRA, body shape of the patient with or without a bustier corset will be captured with a handheld 3D scanner and input into a 3D printer for PERSBRA design and manufacturing. A participant will receive two more CT scans in addition to the simulation scan with PERSBRA in place before the first and the sixth fractions of irradiation. These images will be analyzed for dosimetric parameters in the presence/absence of PERSBRA as well as position reproducibility. The data will provide proof-of-principle evidence for the clinical utility of PERSBRA and will facilitate its further refinement.

DETAILED DESCRIPTION:
1. Patients with early breast cancer or ductal carcinoma in situ treated with breast conservation surgery.
2. Adjuvant radiotherapy to the breast is part of the patient's initial treatment plan.
3. Non-contrast CT scan is a routine procedure for the patient's radiotherapy treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early breast cancer or carcinoma in situ after partial mastectomy have decided to receive adjuvant radiation therapy for the breast on the affected side, and use non-contrast computed tomography to obtain localized images is part of the original treatment plan.

Exclusion Criteria:

* Clinical diagnosis or pathological diagnosis has lymph node metastasis, lymph node micrometastasis, or lymph node tumor cells.
* The clinical diagnosis is likely to have metastatic cancer.
* Pregnant women.
* Be younger than 20 years old.
* The subject was unable to read and understand the subject consent form written in Chinese and complete the informed consent procedure.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-04-21 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Irradiated cardiac dose | Time Frame: At simulation, expected average of 1 week
  Radiation dose distribution of the cardiopulmonary on the affected side.

SECONDARY OUTCOMES:
Irradiated dose of left anterior descending artery | Time Frame: At simulation, expected average of 1 week
  Radiation dose distribution of the left anterior descending artery on the affected side.
Irradiated lung dose | At simulation, expected average of 1 week
  Radiation dose distribution of the lung on the affected side.
Clinical target volume | At simulation, expected average of 1 week
  Radiation dose distribution of clinical target volume.
Irradiated dose of axillary lymphatic area | At simulation, expected average of 1 week
  Irradiated dose of axillary lymphatic area.

CONTACTS AND LOCATIONS:
Overall Officials: Long-Sheng Lu, MD, Ph.D., Study Director — Taipei Medical University Hospital; Jeng-Feng Chiou, MD, Ph.D., Study Chair — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whelan TJ, Olivotto IA, Parulekar WR, Ackerman I, Chua BH, Nabid A, Vallis KA, White JR, Rousseau P, Fortin A, Pierce LJ, Manchul L, Chafe S, Nolan MC, Craighead P, Bowen J, McCready DR, Pritchard KI, Gelmon K, Murray Y, Chapman JA, Chen BE, Levine MN; MA.20 Study Investigators. Regional Nodal Irradiation in Early-Stage Breast Cancer. N Engl J Med. 2015 Jul 23;373(4):307-16. doi: 10.1056/NEJMoa1415340. PMID 26200977
- [Background] Poortmans PM, Collette S, Kirkove C, Van Limbergen E, Budach V, Struikmans H, Collette L, Fourquet A, Maingon P, Valli M, De Winter K, Marnitz S, Barillot I, Scandolaro L, Vonk E, Rodenhuis C, Marsiglia H, Weidner N, van Tienhoven G, Glanzmann C, Kuten A, Arriagada R, Bartelink H, Van den Bogaert W; EORTC Radiation Oncology and Breast Cancer Groups. Internal Mammary and Medial Supraclavicular Irradiation in Breast Cancer. N Engl J Med. 2015 Jul 23;373(4):317-27. doi: 10.1056/NEJMoa1415369. PMID 26200978
- [Background] Deasy JO, Bentzen SM, Jackson A, Ten Haken RK, Yorke ED, Constine LS, Sharma A, Marks LB. Improving normal tissue complication probability models: the need to adopt a "data-pooling" culture. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3 Suppl):S151-4. doi: 10.1016/j.ijrobp.2009.06.094. PMID 20171511
- [Background] Formenti SC, DeWyngaert JK, Jozsef G, Goldberg JD. Prone vs supine positioning for breast cancer radiotherapy. JAMA. 2012 Sep 5;308(9):861-3. doi: 10.1001/2012.jama.10759. No abstract available. PMID 22948692
- [Background] Bruzzaniti V, Abate A, Pinnaro P, D'Andrea M, Infusino E, Landoni V, Soriani A, Giordano C, Ferraro A, Strigari L. Dosimetric and clinical advantages of deep inspiration breath-hold (DIBH) during radiotherapy of breast cancer. J Exp Clin Cancer Res. 2013 Nov 7;32(1):88. doi: 10.1186/1756-9966-32-88. PMID 24423396
- [Background] Moon SH, Shin KH, Kim TH, Yoon M, Park S, Lee DH, Kim JW, Kim DW, Park SY, Cho KH. Dosimetric comparison of four different external beam partial breast irradiation techniques: three-dimensional conformal radiotherapy, intensity-modulated radiotherapy, helical tomotherapy, and proton beam therapy. Radiother Oncol. 2009 Jan;90(1):66-73. doi: 10.1016/j.radonc.2008.09.027. Epub 2008 Nov 5. PMID 18992950

DOCUMENTS (1):
  • Informed Consent Form (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT04929197/ICF_000.pdf